CLINICAL TRIAL: NCT02661516
Title: Clinical and Economic Burden of Bleeding Events in Patients in the UK With Non-Valvular Atrial Fibrillation Treated With Vitamin K Antagonists
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV185-338
Record Dates: First submitted 2016-01-19; First posted 2016-01-22 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Vitamin K Antagonists: Vitamin K Antagonists dose as specified

SUMMARY:
The purpose of the study is to estimate the impact of bleeding events in patients in the UK with non-valvular atrial fibrillation (NVAF) treated with vitamin K antagonists (VKA).

ELIGIBILITY:
Inclusion Criteria:-

For the CPRD-HES cohort, patients will be included if they meet these criteria:

* Have CPRD data linked to HES
* Have an AF diagnosis (based on Read codes from CPRD or ICD-10 codes from HES) and have been treated with VKA during the study period

  -≥18 years old at index date
* CPRD acceptability quality criteria are present.

For the CPRD cohort, patients will be included if they meet the following criteria:

* Have an Atrial Fibrillation (AF) diagnosis (based on Read codes from CPRD) and have been treated with VKAs during the study period
* ≥18 years old at index date
* CPRD acceptability quality criteria are present.

Exclusion Criteria:

For the two cohorts of interest, patients will be excluded if they meet the following criteria:

* Fewer than 12 months of computerised data available prior to the index date (in order to provide a minimum amount of computerised history and to avoid issues associated with updating records when a patient joins a practice). The date of start of computerized records will be the latter of the patient's date of registration with the practice or the practice's Up-to-Standard (UTS) date (when the practice is deemed to be contributing data of adequate quality)
* The practice is not UTS, or the patient is deemed "unacceptable" according to CPRD's quality criteria
* There is evidence of valvular disease, repair, or replacement before (ie, up to 12 months prior to the index date) or during the study period
* There are records of Novel anticoagulant (NOAC)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective cohort with study period from January 1, 2003 to December 31, 2013 using the Clinical Practice Research Datalink (CPRD). The study will identify AF patients treated with VKA during the study period and will follow them from the first record of VKA use (index date). until the first of end of study period, leaving the database, VKA discontinuation/switch, or death. It will use person-time denominators to handle the varying length of follow-up of patients
Sampling Method: Non-Probability Sample
Enrollment: 16513 (Actual)
Dates: Start 2014-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Impact of bleeding events on the risk of subsequent clinical events including subsequent bleeds assessed based on hazard ratios | Up to 24 months after initial treatment with VKA
Impact of bleeding events on the rate of health-care resource utilization (HCRU) assessed based on incidence rate ratios | Up to 24 months after initial treatment with VKA
Impact of bleeding events on the health-care costs in NVAF patients treated by VKAs assessed based on ratios of costs associated with number of bleeding events | Up to 24 months after initial treatment with VKA

SECONDARY OUTCOMES:
Variation of impact of bleeding events on clinical events, the rate of HCRU, and health-care costs over time following each bleeding event in NVAF patients treated by VKA | Upto 24 months after initial treatment with VKA
Characteristics of NVAF patients newly treated with VKA who experience bleeding events | Up to 24 months after initial treatment with VKA
Characteristics of NVAF patients newly treated with VKA who do not experience bleeding events | Up to 24 months after initial treatment with VKA

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx